CLINICAL TRIAL: NCT00004568
Title: Clinical and Molecular Manifestations of Inherited Neurological Disorders
Brief Title: Study of Inherited Neurological Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000043; 00-N-0043
Record Dates: First submitted 2000-02-11; First posted 2000-02-14 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11-06

CONDITIONS: Motor Neuron Disease; Muscular Disease; Muscular Dystrophy; Peripheral Nervous System Disease
Keywords: Myopathy; Muscular Dystrophy; Motor Neuron Disease
MeSH Terms: conditions — Motor Neuron Disease; Muscular Diseases; Muscular Dystrophies; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inherited Neurological Patients: Includes individuals and families with a known or unknown inherited neurological condition.

SUMMARY:
This study is designed to learn more about the natural history of inherited neurological disorders and the role of heredity in their development. It will examine the genetics, symptoms, disease progression, treatment, and psychological and behavioral impact of diseases in the following categories: hereditary peripheral neuropathies; hereditary myopathies; muscular dystrophies; hereditary motor neuron disorders; mitochondrial myopathies; hereditary neurocognitive disorders; inherited neurological disorders without known diagnosis; and others. Many of these diseases, which affect the brain, spinal cord, muscles, and nerves, are rare and poorly understood.

Children and adults of all ages with various inherited neurological disorders may be eligible for this study. Participants will undergo a detailed medical and family history, and a family tree will be drawn. They will also have a physical and neurological examination that may include blood test and urine tests, an EEG (brain wave recordings), psychological tests, and speech and language and rehabilitation evaluations. A blood sample or skin biopsy may be taken for genetic testing. Depending on the individual patient s symptoms, imaging tests such as X-rays, CT or MRI scans and muscle and nerve testing may also be done.

Information from this study may provide a better understanding of the genetic underpinnings of these disorders, contributing to improved diagnosis, treatment, and genetic counseling, and perhaps leading to additional studies in these areas.

DETAILED DESCRIPTION:
The Neurogenetics Branch (NGB) within the National Institute of Neurological Disorders and Stroke (NINDS) is conducting a study to evaluate and provide genetic diagnosis to participants with various diagnosed and undiagnosed neurological conditions.

OBJECTIVES:

The primary objective of this protocol is to provide a resource of participants for enrollment into new research protocols throughout the NGB and other NIH laboratories. Evaluating and diagnosing participants will allow the NGB specialists to maintain their expertise and gain additional knowledge of the course of various neurological disorders. The information obtained will allow for the evaluation and diagnosis of the studied neurological diseases. This understanding may lead to ideas for future protocols. In some cases, blood or other biologic samples (including urine, saliva, or a cheek (buccal) swab) will be obtained for future laboratory studies.

STUDY POPULATION

The number of participants to be enrolled will be set to 3,500 participants with neurological diseases and their unaffected relatives.

DESIGN:

This is an observational diagnostic study of multiple neurological diseases and their pathophysiology.

OUTCOME MEASURES:

No formal outcomes will be measured; however the clinical assessments of enrolled participants can be used to characterize the disease manifestations. In addition, DNA samples obtained may be used to identify and verify causative mutations as well as identify novel genes, which may help establish pathogenic mechanisms and genotype-phenotype correlations.

ELIGIBILITY:
* Participants include those with inherited neurological conditions based on the training and research needs of the Neurogenetics Branch program. There is no logical limit; however the total number of participants that can be enrolled in the protocol will be restricted. No more than 3,500 participants with either diagnosed or undiagnosed neurological conditions and their unaffected relatives will be enrolled in this evaluation and diagnostic protocol.

INCLUSION CRITERIA:

Participants will be eligible if they:

* Have either a known or suspected, inherited neurological disease, OR are an unaffected relative (first-, second-, third, or higher degree relative) of a participant with a genetic neurological disease.
* Have the ability to understand and sign an informed consent or have a parent/legal guardian to do so if they are minor children or a legal guardian to provide consent for adults without consent capacity.
* Aged 2 years and above.

EXCLUSION CRITERIA:

Participants will not be eligible if they:

-Have a systemic disease that compromises the ability to provide adequate neurologic examination or diagnosis.An example of this would be a contagious disease that would compromise our ability to do an adequate neurological exam.

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: general population
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2000-02-18 (Actual)

PRIMARY OUTCOMES:
Genetic disease identification; Deep phenotyping of rare genetic neurological disorders; Training of fellows and students | Outcome measures assessed at initial visit and ongoing until a genetic diagnosis is made. Duration of study 15 years (per protocol).
  The primary objective of this protocol is to provide a resource of participants for enrollment into new research protocols throughout the NGB and other NIH laboratories. Evaluating and diagnosing participants will allow the NGB specialists to maintain their expertise and gain additional knowledge of the course of various neurological disorders. The information obtained will allow for the evaluation and diagnosis of the studied neurological diseases. This understanding may lead to ideas for future protocols. In some cases, blood or other biologic samples (including urine, saliva, or a cheek (buccal) swab) will be obtained for future laboratory studies. No formal outcomes will be measured; however, the clinical assessments of enrolled participants can be used to characterize the disease manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Grunseich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (2):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- University of Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-N-0043.html